CLINICAL TRIAL: NCT06266182
Title: The Effect of an Online Acceptance and Commitment Intervention on Meaning-Making Process in Cancer Patients Following Hematopoietic Cell Transplantation: a Randomized Controlled Trial Enhanced With a Single-case Experimental Design
Brief Title: The Effect of an Online ACT Intervention on Meaning-Making Process in Cancer Patients Following Hematopoietic Cell Transplantation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Social Sciences and Humanities, Warsaw (Other)
Collaborators: National Science Centre, Poland (Other Government)
Responsible Party: Principal Investigator, Aleksandra Kroemeke, PhD, Associate professor, University of Social Sciences and Humanities, Warsaw
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2020/39/B/HS6/01927
Record Dates: First submitted 2024-01-25; First posted 2024-02-20 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Hematopoietic Cell Transplantation Recipient; Acceptance and Commitment Therapy
Keywords: cancer patients; hematopoietic cell transplantation; ACT-based intervention; web-based intervention; meaning-making; subjective well-being; psychological flexibility; randomized controlled trial; single-case experimental design
MeSH Terms: interventions — Acceptance and Commitment Therapy; Educational Status

STUDY DESIGN:
Intervention Model Description: This trial is enhanced by a single-case experimental design (SCED), in which all study participants will receive the same intervention (i.e., intervention study model: single group). In SCED, there is no masking. The estimated total number of participants to be enrolled in SCED is 6-9.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACT intervention (Experimental): Participants in the ACT intervention arm will learn new adaptive ways to cope with difficulties (including difficult thoughts or feelings).
  Interventions: Behavioral: Acceptance and Commitment Therapy
- Education (Other): Participants in the Education arm will become familiar with post-HCT recommendations. This will be a minimally enhanced usual care.
  Interventions: Behavioral: Education

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy — ACT intervention will start on the second day after hospital discharge and will take 14 days (+ day 0 with organizational information). Each day, participants will receive a web-based intervention consisting of educational and practical tasks/activities. Participants will learn to recognize moments of choice (actions that lead towards values or away from them) and to use attention flexibly to free themselves from the power of thoughts, to open up and accept emotions, and to be able to determine what is important and take action in line with values. All of the tasks will be available in written form and audio. The ACT intervention is built from standard ACT exercises.
  Other Names: ACT-based intervention; ACT
  Arms: ACT intervention
Behavioral: Education — Education will start on the second day after hospital discharge and will take 14 days (+ day 0 with organizational information). Each day, participants will receive information about post-transplant prescriptions along with exercises to support the implementation. Participants will learn about nutrition, personal hygiene, preventing infections, coping with fatigue, resuming activity, rest and sleep, engaging in social interactions, and sexual health. The content is prepared based on available guides for HCT recipients.
  Arms: Education

SUMMARY:
This trial aimed to test internet-based Acceptance and Commitment Therapy (ACT) intervention to induce a meaning-making process in cancer patients following hematopoietic cell transplantation (HCT). ACT includes identifying personal values and engaging in activities consistent with these values, developing acceptance, as well as focusing on the present moment or performing activities with greater awareness. In total, 192 patients following the first (autologous or allogeneic) HCT will be randomly assigned in equal numbers to either the ACT intervention or an education session. Participants in both conditions will take part in 14-day training (about 5-10 minutes a day). The outcomes will be measured at baseline, during the intervention, immediately, 1 month, and 3 months after the intervention. Moreover, 6-9 additional participants will be randomly assigned to pre-intervention measurement length (1-3 weeks) before completing ACT intervention, followed by 7-day observations at the 2nd and 3rd post-intervention measure. The researchers hypothesized that ACT intervention would foster a meaning-making process and thus reduce distress induced by the discrepancy between global and situational meaning as compared to education.

DETAILED DESCRIPTION:
This trial evaluates the feasibility, acceptability, and preliminary efficacy of self-help internet-based Acceptance and Commitment Therapy (ACT) intervention on meaning-related distress as well as secondary outcomes in patients following hematopoietic cell transplantation (HCT). Randomized controlled trial (RCT) will be enhanced with a single-case experimental design (SCED).

Recruitment will take place at a single center, after elective admission to the bone marrow transplantation and oncohematology unit due to HCT before the start of conditioning treatment. Recruitment will take place on average on the 2nd day after admission. Every two days, the transplant coordinator and physician (members of the research team) will review the lists of patients enrolled for HCT. Those who meet the inclusion criteria will be initially informed of the purpose of the study and invited for an extensive briefing by a recruiter (member of the research team). Patients will also be allowed to ask any remaining questions about the aim of the study and the study procedures. After receiving an extensive briefing, all patients who give written informed consent will proceed with baseline. Data will be collected via a self-reported survey on a mobile device. Clinical data will be obtained from the medical records. All participants will receive written user instructions for the daily sessions and measurements.

In RCT, participants will be randomly assigned in a double-blinded manner to ACT intervention and education conditions at a ratio of 1:1 by a trial coordinator (member of the research team). Randomization will be stratified by type of transplant. Participants and researchers analyzing data will be blind to the allocation of the participants to the conditions. Participants allocated to the ACT intervention will receive online ACT-based intervention within 14 days after hospital discharge. Each day's intervention will consist of an educational and practical part (standard ACT activity) followed by a debrief. On some days, participants will also receive additional exercise (optional). The whole intervention will be tailored to the context of the disease and treatment. During the same period, participants allocated to the education will receive an online guide to post-HCT recommendations. The intervention/education will be discontinued by participants at any time without any negative consequences. During the intervention/education, participants will fill in a short questionnaire assessing potential mediator variables each day, at the beginning of every online session. Participants will receive daily reminders about the intervention/education. Also, direct technical support will be available 24/7. If participants fail to complete study assessments, motivational reminders will be sent by email. If participants drop out or stop using the intervention, they will be asked for the reason(s) why they decided to quit the intervention and/or study.

In SCED, all participants will take part in the online ACT intervention and daily surveys at the 2nd and 3rd post-intervention assessments.

Feasibility will be examined via attrition and adherence rates, as well as questions about intervention engagement. Acceptability will be measured by intervention satisfaction and evaluation (attractiveness and easiness).

ELIGIBILITY:
Inclusion Criteria:

* Qualification for the first autologous or allogeneic HCT due to hematologic malignancies or solid tumors
* Age ≥ 18 years
* Signed written informed consent
* Ability to read and write in Polish
* Daily access to the Internet by computer and/or mobile device

Exclusion Criteria:

* Major psychiatric or cognitive disorder that would impede providing informed consent and study participation
* Inability to cooperate and give informed consent
* Hearing, seeing, or movement impairment that precludes participation
* Current participation in any form of psychotherapy
* No access to the Internet
* No access to a computer and/or mobile device
* Inability to use a computer and/or mobile device and the Internet

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2024-03-06 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Distress (Global Meaning Violation Scale; GMVS) | Change from baseline to immediately, 1 month and 3 months after intervention
  The GMVS measures meaning-related distress. It is a 12-item questionnaire (from the original, the item "health" was removed due to the context of the study) that assesses belief (5 items) and goal violations (7 items) in response to stressors on a 5-point scale ranging from 1 (not at all) to 5 (very much). The overall score is calculated by summing the scores of all 12 items, with a possible range of 12-60. Higher scores indicate greater meaning-related distress (greater global meaning violation).

SECONDARY OUTCOMES:
Illness perception (Brief-Illness Perception Questionnaire; B-IPQ) | Change from baseline to immediately, 1 month and 3 months after intervention
  The B-IPQ measures cognitive and emotional representations of illness. It is an 8-item questionnaire that assesses cognitive illness representation, emotional illness representation, and illness comprehensibility representation on a 0-10 point scale. The total score is calculated by summing the scores of all 8 items, with a possible range of 0-80. Higher scores indicate more threatening perception of the illness.
Global meaning (Meaning in Life Questionnaire; MLQ) | Change from baseline to immediately, 1 month and 3 months after intervention
  The MLQ measures meaning in life. It is a 10-item questionnaire that assesses the Presence of meaning in life and the Searches for meaning in life on a 7-point scale ranging from 1 (absolutely untrue) to 7 (absolutely true). The subscale scores are calculated by summing the scores of relevant items (5 per subscale), with a possible range of 5-35. Higher scores indicate a greater Presence of meaning in life and Search for meaning in life, respectively.
Psychological flexibility (Comprehensive Assessment of Acceptance and Commitment Therapy Processes-9; CompACT-9) | Change from baseline to immediately, 1 month and 3 months after intervention
  The CompACT-9 measures psychological flexibility. It is a 9-item questionnaire that assesses Openness to Experience, Behavioral Awareness, and Valued Action on a 7-point scale ranging from 0 (strongly disagree) to 6 (strongly agree). The overall score is calculated by summing the scores of all 9 items, with a possible range of 0-36. Higher scores indicate higher psychological flexibility (greater openness to experience and willingness to experience internal events such as thoughts, feelings, sensations, etc. without trying to control or avoid them; greater behavioral awareness and mindful attention to current actions; greater engagement in valued actions and meaningful activity).
Coping self-efficacy (Coping Self-Efficacy Scale; CSE - selected items) | Change from baseline to immediately, 1 month and 3 months after intervention
  The CSE measures a perceived self-efficacy for coping with challenges and threats. This study used 6 items tailored to the context of the study (2 per subscale: Problem-focused Coping, Emotion-focused Coping, and Social Support Coping) assessed on a 5-point scale ranging from 1 (not at all) to 5 (strongly). The overall score is calculated by summing the scores of all 6 items, with a possible range of 6-30. Higher scores indicate greater coping self-efficacy.
Deliberate meaning-making (Core Beliefs Inventory; CBI) | Change from baseline to immediately, 1 month and 3 months after intervention
  The CBI is a 10-item questionnaire that assesses deliberate meaning-making coping on a 6-point scale ranging from 0 (not at all) to 5 (to a very degree). The total score is calculated by summing the scores of all 10 items, with a possible range of 0-45. Higher scores indicate greater deliberate searching for meaning.
Automatic meaning-making (Event-Related Rumination Inventory; ERRI - intrusive ruminations subscale) | Change from baseline to immediately, 1 month and 3 months after intervention
  The intrusive ruminations subscale of the ERRI measures automatic meaning-making coping. It is a 10-item subscale that assesses intrusive ruminations on a 4-point scale ranging from 0 (not at all) to 3 (often). The total score is calculated by summing the scores of all 10 items, with a possible range of 0-30. Higher scores indicate greater automatic searching for meaning.
Post-traumatic growth (the "current standing" Post-Traumatic Growth Inventory-Short Form; C-PTGI-SF ) | Change from baseline to immediately, 1 month and 3 months after intervention
  The C-PTGI-SF measures psychological well-being in cross-sectional assessment, as well as posttraumatic growth (element of meanings made) in multiple assessments. It is a 10-item questionnaire that assesses psychological well-being on a 6-point scale ranging from 0 (not at all) to 5 (to a very great degree). The total score is calculated by summing the scores of all 10 items, with a possible range of 0-50. Higher scores indicate better well-being.
Meanings made (Meaning of Loss Codebook; MLC) | Change from baseline to immediately, 1 month and 3 months after intervention
  The MLC evaluates meanings made. It is a 3-item tool that assesses sense made, benefit finding, and sense of identity change on a 5-point scale ranging from 1 (not at all) to 5 (to a very great degree). The overall score is calculated by summing the scores of all 3 items, with a possible range of 3-15. Higher scores indicate greater meanings made.
Anxiety and depressive symptoms (Patient Health Questionnaire-4; PHQ-4) | Change from baseline to immediately, 1 month and 3 months after intervention
  The PHQ-4 is a 4-item questionnaire that assesses symptoms of anxiety (2 items) and depression (2 items) on a 4-point scale ranging from 0 (not at all) to 3 (nearly every day). The subscale scores are calculated by summing the scores of 2 items, with a possible range of 0-6. Higher scores indicate higher levels of anxiety and depression symptoms, respectively. The total PHQ-4 score complements the subscale scores as an overall measure of symptom burden, as well as functional impairment and disability.
Loneliness (The Revised UCLA Loneliness Scale; R-UCLA - selected items) | Change from baseline to immediately, 1 month and 3 months after intervention
  The R-UCLA measures perceived social isolation. This study used 5 items that assess the emotional and social aspects of loneliness on a 4-point scale ranging from 1 (never) to 4 (often or always). The total score is calculated by summing the scores of all 5 items, with a possible range of 5-20. Higher scores indicate greater loneliness.
Loneliness (the Community Life Survey) | Change from baseline to immediately, 1 month and 3 months after intervention
  A direct question about loneliness from the Community Life Survey is used. The statement is assessed on a 4-point scale ranging from 1 (never) to 4 (often or always). A higher score indicates greater loneliness.
Health-related quality of life (Quality of Life Questionnaire of the European Organization for Research and Treatment of Cancer; EORTC QLQ-C3) | Change from baseline to immediately, 1 month and 3 months after intervention
  The EORTC QLQ-C30 measures the health-related quality of life of cancer patients. It is a 30-item questionnaire that assesses physical, role, social, emotional, and cognitive functioning, as well as various symptoms, financial impact, and global quality of life. Twenty-eight items are rated on a 4-point scale ranging from 1 (not at all) to 4 (very much), while 2 items are rated on a 7-point scale ranging from 1 (very poor) to 7 (excellent). The overall score is calculated by summing the scores of all items, with a possible range of 0-100. Higher scores indicate better function and a higher quality of life.
Daily subjective health (Daily Subjective Health Scale) | RCT: day-by-dy for 14 days during the intervention. SCED: for 7-21 days before intervention, day-by-dy for 14 days during the intervention, for 7 days immediately, 1 month, and 3 months after intervention
  Daily subjective health is measured by a single-item statement "Generally, I can say my health today was …" on a 5-point scale ranging from 1 (bad) to 5 (excellent). Higher scores indicate greater daily physical health.
Daily affect (Daily Positive and Negative Affect Scale) | RCT: day-by-dy for 14 days during the intervention. SCED: for 7-21 days before intervention, day-by-dy for 14 days during the intervention, for 7 days immediately, 1 month, and 3 months after intervention
  The Daily Positive and Negative Affect Scale is a 4-item questionnaire that consists of two positive (happy, cheerful) and two negative adjectives (sad, gloomy) rated on a 5-point scale ranging from 1 (not at all) to 5 (to a very great degree). The subscale scores are calculated by summing the scores of relevant items, with a possible range of 2-10. Higher scores indicate higher daily positive or negative affect.
Daily meaning-making (Event-Related Rumination Inventory-daily form; ERRI-daily form) | RCT: day-by-dy for 14 days during the intervention. SCED: for 7-21 days before intervention, day-by-dy for 14 days during the intervention, for 7 days immediately, 1 month, and 3 months after intervention
  The ERRI-daily form measures deliberate and automatic meaning-making coping. It is a 4-item tool that assesses deliberate and intrusive ruminations on a 4-point scale ranging from 0 (not at all) to 3 (to a very great degree). The subscale scores are calculated by summing the scores of relevant items (2 per subscale), with a possible range of 0-6. Higher scores indicate greater deliberate or automatic searching for meaning.
Daily meanings made (Meaning of Loss Codebook-daily form; MCL-daily form) | RCT: day-by-dy for 14 days during the intervention. SCED: for 7-21 days before intervention, day-by-dy for 14 days during the intervention, for 7 days immediately, 1 month, and 3 months after intervention
  The MLC-daily form measures daily meanings made. It is a 3-item tool that assesses daily sense made, benefit finding, and sense of identity change on a 5-point scale ranging from 1 (not at all) to 5 (to a very great degree). The overall score is calculated by summing the scores of all 3 items, with a possible range of 3-15. Higher scores indicate greater daily meanings made.
Daily psychological flexibility (Comprehensive Assessment of Acceptance and Commitment Therapy Processes-daily form; CompACT-daily form) | RCT: day-by-dy for 14 days during the intervention. SCED: for 7-21 days before intervention, day-by-dy for 14 days during the intervention, for 7 days immediately, 1 month, and 3 months after intervention
  The CompACT-daily form is a 4-item tool that assesses daily psychological flexibility (i.e. daily Openness to experience - 2 items, daily Behavioral awareness - 1 item, and daily Valued action - 1 item) on a 7-point scale ranging from 0 (strongly disagree) to 6 (strongly agree). The overall score is calculated by summing the scores of all 4 items, with a possible range of 0-24. Higher scores indicate higher daily psychological flexibility (i.e. greater daily openness to experience and willingness to experience internal events such as thoughts, feelings, sensations, etc. without trying to control or avoid them; greater daily behavioral awareness and mindful attention to current actions; greater daily engagement in valued actions and meaningful activity).

CONTACTS AND LOCATIONS:
Overall Officials: Aleksandra Kroemeke, PhD, Principal Investigator — SWPS University (University of Social Sciences and Humanities)
Locations (1):
- Maria Skłodowska-Curie National Research Institute of Oncology Gliwice Branch, Department of Bone Marrow Transplantation and Oncohematology, Gliwice, Poland

IPD SHARING:
Plan to Share IPD: Yes
The full protocol, dataset, statistical codes, and outputs will be made available at the Open Science Framework (OSF). Anonymized participant-level datasets will be publicly available, however, without demographics and clinical data due to privacy or ethical restrictions (the possibility of identification of participants).
  The data will be stored for at least 5 years after the end of the project unless other regulations lengthen the need to store the data or it is not necessary due to other reasons (e.g. documentation of research results).
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Beginning 3 months after publication without an end date.
Access Criteria: All those who will have an open link.
URL: https://osf.io/hxfsg

REFERENCES:
- [Derived] Kroemeke A, Dudek J, Kijowska M, Owen R, Sobczyk-Kruszelnicka M. The effect of an online acceptance and commitment intervention on the meaning-making process in cancer patients following hematopoietic cell transplantation: study protocol for a randomized controlled trial enhanced with single-case experimental design. Trials. 2024 Jun 18;25(1):392. doi: 10.1186/s13063-024-08235-1. PMID 38890709